CLINICAL TRIAL: NCT07127835
Title: Provocation After Nurse-Directed Assessment (PANDA) Study
Acronym: PANDAS
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Prof., The University of Hong Kong
Other Study IDs: PANDAstudy
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Drug Allergy; Penicillin Allergy
Keywords: Nurse-led Service; Drug Provocation Test; Delabelling
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurse-led group: Receive Nurse-led penicillin allergy delabelling service
  Interventions: Diagnostic Test: Nurse-led penicillin allergy delabelling service
- Allergist-led group: Receive Allergist-led penicillin allergy delabelling service
  Interventions: Diagnostic Test: Allergist-led penicillin allergy delabelling service

INTERVENTIONS:
Diagnostic Test: Nurse-led penicillin allergy delabelling service — Patients in this group undergo risk assessment and categorization by nurses to identify low-risk individuals for delabeling. For these patients, nurses will collaborate with allergists in the delabeling process.
  Groups: Nurse-led group
Diagnostic Test: Allergist-led penicillin allergy delabelling service — Patients assigned to this group will undergo risk assessment and delabeling led by allergists for both low-risk and high-risk cases.
  Groups: Allergist-led group

SUMMARY:
The study aims to evaluate the effectiveness and safety of a collaborative nurse-allergist approach in penicillin allergy delabeling services. It also seeks to assess the impact on patients' quality of life and compare resource utilization and cost-effectiveness between the nurse-allergist collaborative approach and the traditional allergist-led approach.

DETAILED DESCRIPTION:
This study hypothesizes that by involving both nurses and allergists in the delabeling process and categorizing patients based on risk levels, it will achieve comparable success rates, safety, and improvements in patients' quality of life. This approach is expected to offer superior advantages in terms of time efficiency, resource utilization, and cost-effectiveness compared to traditional allergist-led services.

ELIGIBILITY:
Inclusion Criteria:

* Receiving inpatient or outpatient treatment at a participating hospital during the study period;
* Possessing a documented penicillin allergy label;
* Underwent penicillin allergy evaluation by the nurse-allergist collaborative approach or the traditional allergist-led approach
* Demographic and clinical data required for the study available.

Exclusion Criteria:

* Patients unable to provide a complete medication history or history of penicillin allergy;
* Patients with only emergency or short-term treatment records;
* Patients who have taken steroids, antihistamines, or similar medications within the last 3 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at a participating hospital who have a documented penicillin allergy label, are evaluated for penicillin allergy through either the nurse-allergist or allergist-led approach, and have available demographic and clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Delabelling Success Rate | 6 months
  Assess the proportion of low-risk patients who are no longer considered allergic to penicillin after delabeling.

SECONDARY OUTCOMES:
Health-Related Quality of Life | 6 months
  Measure changes in patients' quality of life before and after delabeling using the validated Drug Hypersensitivity Quality of Life Questionnaire (DrHy-Q). The DrHy-Q is a 15-item instrument answered on a 5-point Likert scale, with scores ranging from 15 (no QoL impairment) to 225 (worst QoL impairment).
Antibiotic Usage Rate | 6 months
  Evaluate changes in the usage rates of penicillin and alternative antibiotics after delabeling.
Age Group Analysis | 6 months
  Compare delabeling success rates across different age groups (e.g., 18-30 years, 31-50 years, and 51 years and older).
Immunocompetence Status | 6 months
  Analyze differences in delabeling success rates and safety between immunocompetent and immunocompromised patients.
Initial vs. Recurrent Labeling | 6 months
  Compare delabeling success rates between patients with an initial penicillin allergy label and those with recurrent labels.

CONTACTS AND LOCATIONS:
Locations (4):
- Hong Kong (4):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schnyder B, Pichler WJ. Mechanisms of drug-induced allergy. Mayo Clin Proc. 2009 Mar;84(3):268-72. doi: 10.4065/84.3.268. PMID 19252115
- [Background] Abrams EM, Khan DA. Diagnosing and managing drug allergy. CMAJ. 2018 Apr 30;190(17):E532-E538. doi: 10.1503/cmaj.171315. No abstract available. PMID 29712672
- [Background] Classen DC, Pestotnik SL, Evans RS, Lloyd JF, Burke JP. Adverse drug events in hospitalized patients. Excess length of stay, extra costs, and attributable mortality. JAMA. 1997 Jan 22-29;277(4):301-6. PMID 9002492
- [Background] Pourpak Z, Fazlollahi MR, Fattahi F. Understanding adverse drug reactions and drug allergies: principles, diagnosis and treatment aspects. Recent Pat Inflamm Allergy Drug Discov. 2008 Jan;2(1):24-46. doi: 10.2174/187221308783399289. PMID 19075990
- [Background] Patton K, Borshoff DC. Adverse drug reactions. Anaesthesia. 2018 Jan;73 Suppl 1:76-84. doi: 10.1111/anae.14143. PMID 29313907